CLINICAL TRIAL: NCT02098200
Title: Percutaneous Treatment of Tricuspid Valve Regurgitation With the TriCinch System™
Acronym: PREVENT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4Tech Cardio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PREVENT_001/2013
Record Dates: First submitted 2014-03-13; First posted 2014-03-27 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Tricuspid Regurgitation
Keywords: tricuspid; regurgitation; repair; outcomes
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Percutaneous treatment of TR by TriCinch (Experimental): Percutaneous treatment of Tricuspid Regurgitation with TriCinch System
  Interventions: Device: TriCinch System

INTERVENTIONS:
Device: TriCinch System — Percutaneous treatment of Tricuspid Regurgitation

SUMMARY:
The TriCinch System™ is intended for percutaneous treatment of tricuspid regurgitation.

It is a percutaneous catheter-based device designed for tricuspid valve repair in order to decrease effective cross-sectional area and relieve symptoms in patients with tricuspid valve regurgitation.

DETAILED DESCRIPTION:
Implantation Procedure: Unlike the standard open chest, arrested heart approach, the 4TECH TriCinch System™ provides a percutaneous solution for tricuspid valve regurgitation treatment: this procedure is performed through deep sedation, while the heart is beating, without the need for respiratory assistance.

The TriCinch System™ consists of a Delivery System that enables transcatheter placement of an implant that can be adjusted to correct Tricuspid valve regurgitation. The TriCinch Delivery System is inserted from the femoral vein to access the right atrium of the heart. At the end of the correction process, the TriCinch Delivery System and the venous introducer are removed and the procedure is concluded.

ELIGIBILITY:
Inclusion Criteria:

* Functional symptomatic tricuspid regurgitation (TR) 2+ to 4+ on a scale of 4+ (moderate to severe), with annular dilatation greater than 40mm.
* Signed informed consent form prior to any study-related procedure.
* Available and able to return to the study site for post-procedural follow-up examination
* Eighteen (18) years of age or older.

Exclusion Criteria:

* Requirement for concomitant cardiac procedure (other than atrial fibrillation correction surgery, closure of PFO (Patent Foramen Ovale) or ASD (Atrial Septal Defect), or PTCA (percutaneous treatment of coronary artery) or CAD (coronary artery bypass surgery) from 1 to 3 months after or before other procedure.
* Presence of any known life threatening (non-cardiac major or progressive disease), non-cardiac disease that will limit the subject's life expectancy to less than one year.
* Cerebro-vascular event within the past 6 months.
* History of mitral/tricuspid endocarditis within the last 12 months.
* Organic tricuspid disease.
* Contraindication or known allergy to device's components, aspirin, anti-coagulation therapy or contrast media that cannot be adequately premeditated.
* Severe hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg, measurement done by sphygmomanometer with stethoscope, allow the patient to sit for at least 5 minutes before beginning BP measurements).
* Female patient is pregnant (urine HCG test result positive) or lactating.
* Known alcohol or drug abuser.
* Currently participating in the study of an investigational drug or device.
* At heart team's judgement, patient IVC dimension is not adequate for device implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Safety: The percentage of participants with Major Adverse Events within 30 days of the procedure. | Up to 30 days
  Freedom from major adverse event: death, Q-wave myocardial infarction, cardiac tamponade, cardiac surgery for failed TriCinch implantation, stroke, or septicaemia.
Performance: The reduction in degree of tricuspid regurgitation measured immediately after the procedure compared to baseline. | intraoperative
  Ability to reduce tricuspid regurgitation by at least 1 degree immediately following implantation of the TriCinch device assessed by means of quantitative echocardiographic parameters.
Performance: The reduction in the degree of tricuspid regurgitation measured at time of discharge compared to baseline. | Time of discharge - 5 days
  Ability to reduce tricuspid regurgitation by at least 1 degree immediately following implantation of the TriCinch device assessed by means of quantitative echocardiographic parameters.

SECONDARY OUTCOMES:
Safety: The percentage of participants with Major Adverse Events up to 3 months of the procedure. | 3 months
  Rate of device-related major adverse event (MAE).
Safety: The percentage of participants with Major Adverse Events within 6 months of the procedure. | 6 months
  Rate of device-related Major Adverse Event (MAE).
Performance: Assessment in the degree of Tricuspid Regurgitation at 3 months compared to baseline. | 3 months
  Ability to maintain Tricuspid Regurgitation with respect to baseline.
Performance: Assessment in the degree of Tricuspid Regurgitation at 6 months compared to baseline. | 6 months
  Ability to maintain Tricuspid Regurgitation with respect to baseline.

OTHER OUTCOMES:
Quality of Life assessment | 6 months
  Compare to baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — San Raffaele Hospital
Locations (14):
- France (3):
  - Bichat Hospital, Paris, Paris Cedex 18
  - Hospices Civils de Lyon, Lyon
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Universitatsklinikum Bonn, Bonn
  - CardioVasculares Centrum Frankfurt, Frankfurt am Main
  - UKE Heart Center, Hamburg
- Italy (7):
  - Monzino Hospital, Milan, Lombardy
  - University Hospital Pisa, Pisa, Tuscany
  - Ferrarotto Hospital, Catania
  - Fondazione Toscana G. Monasterio Ospedale del Cuore G. Pasquinucci, Massa
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione PTV Policlinico Tor Vergata, Roma
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands